CLINICAL TRIAL: NCT00434720
Title: Comparison of GlideScope Specific Stylet to Malleable Stylet for GlideScope Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Timothy Turkstra, University of Western Ontario
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R-06-490; 12754
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Intubation, Endotracheal
Keywords: GlideScope; Stylet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: GlideScope Specific Stylet

SUMMARY:
The GlideScope video laryngoscope (Verathon) is an intubating device that uses a high-resolution camera embedded into a plastic laryngoscope blade. An LED provides illumination. The GlideScope often provides a good laryngoscopic view, but passing the endotracheal tube (ETT) through the vocal cords is sometimes difficult. Because of the 60 degree anterior curvature of the GlideScope's blade, ETT's must have stylets inserted so that the ETT distal tip can be positioned anteriorly. Various authors have recommended different angles of the ETT to optimally place it into the trachea. Previous study demonstrated that 90 degree sharp bend was both faster and subjectively easier in a heterogeneous group of intubators. With the introduction of a rigid GlideScope Specific Stylet by the manufacturer, the question arises as to the the best configuration of stylet for the ETT. Therefore, this prospective, randomized, single-blinded trial is proposed.

The null hypothesis is that there will be no difference between the GlideScope Specific Stylet and the standard malleable stylet.

DETAILED DESCRIPTION:
Purpose:

To determine the optimum angle of curvature of an endotracheal tube when used with a GlideScope in order to intubate in the most efficient fashion.

Methods:

Groups: A) 90º curvature, malleable stylet B) shallow curvature, rigid GlideScope Specific Stylet

Hypothesis:

The null hypothesis is that there is no difference in the primary outcome (time to intubation). i.e. we hypothesize that the time to intubate is not related to the shape of the endotracheal tube. The control group will be arbitrarily assigned to the 90º group that was the preferred option in a previous trial.

Primary Endpoint:

1) Time to intubation (seconds).

Written informed consent will be obtained by one of the study investigators, and a copy will be given to each participant. Written informed consent will also be obtained from the operator of the GlideScope. After consent, randomization will occur by selecting the next consecutive envelope.

There are three distinct anesthesia providers involved in the conduct of this study, as follows:

1. "operator" - person performing the intubation
2. "timer" - person timing the outcome (one of the co-investigators)
3. "shaper" - person who ensures that the angle and stylet of the tube matches the group to which the patient was allocated

Because the person intubating must be blind up until the time at which the tube is to be used, the unopened envelope will be taken to a third anesthesia provider, who will prepare the ETT with stylet in an area that is not visible to the person performing the intubation or to the person timing the intubation. The person performing the intubation will specify what size of tube they wish to use. This will most commonly be 7.5 mm internal diameter (ID) for a female and 8.0 ID for males, but the operator is free to use whatever size they feel is appropriate. The tube size selection will take place before unblinding so the group allocation cannot affect the decision of tube size.

"Group A" ETT's will be shaped with the aid of a standard malleable stylet (Rusch 14 Fr) that has been lubricated with single-use water-soluble lubricant. "Group B" ETT's will be instrumented with the GlideScope Specific Stylet, with identical lubricant. The prepared tube will then be concealed under a standard green OR towel and brought to the operating room (OR). This tube will be placed close to the patient's head so that it is readily accessible.

Data Collection

In the OR, the GlideScope will be turned on at least 60s before use to prevent fogging. The patient will be cared for in the usual fashion with respect to monitoring and induction of general anesthesia. Muscle relaxation will be used, and the agent used is at the discretion of the operator. After induction of anesthesia, bag-mask ventilation will be used in the usual fashion until the operator decides to proceed to laryngoscopy with the GlideScope. The operator will remain blinded to the group allocation until after the laryngoscopic view has been obtained with the GlideScope, where upon he will be handed the endotracheal tube.

The timer (who cannot see the tube under the green towel) will watch the operator until the GlideScope is in the patient's mouth, start the timer, and then turn 180º to face the anesthetic monitor. The timer will not be able to see the ETT, stylet, or curvature because he will be facing the screen.

Timing will continue until end-tidal CO2 of at least 30 mmHg is seen on the anesthesia monitor, at which point the data collection form will be filled out, and the study protocol will be finished. (The time to intubation will be recorded to the nearest tenth of a second.) If the operator fails to intubate within 3 attempts or 150 seconds, the intubation will be noted as a failure, and the ultimately successful means of securing the airway will be recorded.

If oxygen desaturation (as recorded by pulse oximetry) below 95% occurs, then the patient will be ventilated in the usual fashion to ensure oxygenation, and re-attempting intubation using the GlideScope may proceed, but the timing will continue, and the same limits to successful intubation (within 3 attempts or total of 150s) will apply. Between attempts, the tube may be re-shaped by the operator if a malleable stylet is used and either the original curvature has been lost or the operator feels that another curvature would be preferred.

Discontinuation Criteria

If the oxygen saturation falls below 90% occurs at any point, the protocol will stop immediately, and management will proceed in the normal fashion at the discretion of the attending anesthesiologist, which could involve immediate intubation using the GlideScope or other intubation device, or ventilation using a mask or laryngeal mask airway. If, at any time, the attending anesthesiologist believes there is any risk to the patient because of the study protocol, the protocol will be terminated and normal anesthetic care will continue.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient scheduled for elective surgery.
* ETT is indicated for the procedure in the opinion of the attending anesthesiologist.
* operator who has performed ≥ 10 GlideScope intubations.

Exclusion Criteria:

* GlideScope contraindicated in the opinion of the attending anesthesiologist.
* known cervical spine abnormalities.
* known or probable difficult airways.
* rapid sequence induction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Duration of Intubation | Timed intubation

SECONDARY OUTCOMES:
Operator Satisfaction | Post intubation

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Turkstra, M. Eng, MD, Principal Investigator — University of Western Ontario, London Health Sciences Center
Locations (1):
- London Health Sciences Center, London, Ontario, Canada